CLINICAL TRIAL: NCT03127085
Title: Patient Specific Reasons for Attending the Emergency Department in the Setting of a Background History of Atrial Fibrillation
Brief Title: A.Fib Emergency Department Study Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Principal Investigator, Dr. Benedict Glover, Chief of Cardiac Arrhythmia Service, Queen's University, Kingston, Ontario, Queen's University
Other Study IDs: AF ED
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with a history of atrial fibrillation (AF) who frequently attend the emergency department (ED) with symptoms may not require emergency treatment, and may be more appropriately managed in an alternative outpatient setting. This may be the result of inappropriate or inadequate advice or a lack of patient understanding. The main research objective pertains to the reason for seeking medical attention for AF in the ED, ED management of the patient, outcomes of ED care and alternative strategies.

DETAILED DESCRIPTION:
This study is a multi-centre, multi-provincial, patient survey using mixed methods. 778 patients will be enrolled from 9 centres in 3 provinces from academic, urban, and rural centres to achieve geographical and health system heterogeneity. The planned duration of the entire study (enrollment through follow-up) is approximately 12 months. Patients presenting to the ED with a primary diagnosis of AF and with a prior diagnosis of established AF will be approached to participate. Each centre will be responsible for obtaining local consent. Data will be stored confidentially and securely at the coordinating centre (Queens University, Kingston, Ontario).

Patients who meet the inclusion criteria will be invited to take part at the time of presentation to the ED or after their ED visit. For all enrolled patients, one follow up telephone call will be made within one to four weeks of the ED visit by a social scientist with specialised training in questionnaires based in Queens University, Kingston, Ontario.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Atrial fibrillation is the primary reason for ED visit (documented by 12-lead ECG or Holter rhythm strip by a member of the healthcare team providing care to the patient).
* Patients with an established history of AF (prior diagnosis with ECG / rhythm strip evidence of AF)
* Patient must be literate in English
* Patient must provide informed consent

Exclusion Criteria:

* Male or female < 18 years of age
* Non-English speaking
* unable and/or unwilling to consent
* Acute coronary syndrome (ischemic chest pain, ST changes, + troponin [mild troponin elevation alone does not exclude the patient])
* Cardiogenic shock or class IV congestive heart failure at the time of visit
* Enrolled in a cardiovascular drug or device research study
* New onset atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a known history of atrial fibrillation that seek emergent medical attention for symptoms of atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Patient decisions and perceptions before an after attending the emergency department with symptoms which may be related to atrial fibrillation | All surveys will occur within a time period of less than or equal to four weeks post emergency department visit
  A detailed telephone survey will be performed in which patients with a known history of atrial fibrillation and symptoms which they feel are related to their diagnosis and who are agreeable to take part in the study will be called by a social scientist. They will be asked a series of questions and their responses will be recorded either on a Likert scale (symptom severity, satisfaction with treatment, quality of life) or as qualitative data (exact symptoms, fears and concerns relating to their underlying diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Glover, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre - Kingston General Hospital Site, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong KL, Babiolakis C, Zile B, Bullen M, Haseeb S, Halperin F, Hohl CM, Magee K, Sandhu RK, Tian SY, Kennedy A, Lobban T, Mariano Z, Dorian P, Angaran P, Evans M, Leong-Sit P, Glover BM. Canada-wide mixed methods analysis evaluating the reasons for inappropriate emergency department presentation in patients with a history of atrial fibrillation: the multicentre AF-ED trial. BMJ Open. 2020 Apr 16;10(4):e033482. doi: 10.1136/bmjopen-2019-033482. PMID 32303514